CLINICAL TRIAL: NCT02422524
Title: A Phase I, Single Dose, Open-Label Study Comparing the Pharmacokinetics and Safety of Pretomanid in Subjects With Mild, Moderate, and Severe Hepatic Impairment to Matched, Non-Hepatically Impaired Subjects
Brief Title: Pretomanid in Adults With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The TB hepatic pretomanid PK trial is closed to enrollment. There is no possibility of enrolling and completing the CSR before November 2024.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0053
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2017-12-14

CONDITIONS: Tuberculosis
Keywords: Hepatic; impairment; PA-824; Pharmacokinetics; Safety; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Child-Pugh A (Mild hepatic impairment) (Experimental): 6 Subjects will receive a single oral dose of 200mg Pretomanid tablets on day 1
  Interventions: Drug: PA-824
- Child-Pugh B (Moderate hepatic impairment) (Experimental): 6 Subjects will receive a single oral dose of 200mg Pretomanid tablets on day 1
  Interventions: Drug: PA-824
- Child-Pugh C (Severe hepatic impairment) (Experimental): 6 Subjects will receive a single oral dose of 200mg Pretomanid tablets on day 1
  Interventions: Drug: PA-824
- Non-hepatically impaired controls (Experimental): 18 matched Subjects will receive a single oral dose of 200mg Pretomanid tablets on day 1
  Interventions: Drug: PA-824

INTERVENTIONS:
Drug: PA-824 — Pretomanid (PA-824) is a nitroimidazooxazine. All subjects will receive a single oral dose of 200 mg Pretomanid on day 1.

SUMMARY:
This is a Phase 1, single dose (200 mg), open-label study comparing the pharmacokinetics and safety of Pretomanid in subjects with mild, moderate, and severe hepatic impairment to matched, non-hepatically impaired subjects. There will be approximately 36 total subjects, adult males and females, 18 to 70 years of age, inclusive. The study will be conducted at 2 sites, study duration is approximately 24 months, and subject participation duration is approximately 5 weeks (including screening). Primary objective: To evaluate the pharmacokinetics of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects. Secondary objective: To evaluate the safety of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single dose (200 mg), open-label study comparing the pharmacokinetics and safety of Pretomanid in subjects with mild, moderate, and severe hepatic impairment to matched, non-hepatically impaired subjects. This study will enroll approximately 6 subjects with mild hepatic impairment (Child-Pugh A), approximately 6 subjects with moderate hepatic impairment (Child-Pugh B), approximately 6 subjects with severe hepatic impairment (Child-Pugh C), and approximately 18 matched non-hepatically impaired subjects. Non-hepatically impaired subjects in the control group will be matched to subjects with hepatic impairment based on age (+/- 10 years) and body weight (+/- 20 percent) as measured at screening (Visit 00A). There will be approximately 36 total subjects, adult males and females, 18 to 70 years of age, inclusive. The study will be conducted at 2 sites, study duration is approximately 24 months, and subject participation duration is approximately 5 weeks (including screening). Primary objective: To evaluate the pharmacokinetics of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects. Secondary objective: To evaluate the safety of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Patients with Hepatic Impairment (Groups 1-3):

1. Subject is able to give voluntary written informed consent before any study related procedure is performed.
2. 18-70 years of age, inclusive.
3. Acceptable laboratory values* obtained at screening (within 21 days prior to admission to the confinement/hospital unit) and either at or within 72 hours of admission to the confinement/hospital unit.

   *Chemistry, complete blood count, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), total bilirubin, alkaline phosphatase, albumin, and urinalysis deemed not clinically significant by the investigator.
4. Hepatic impairment classified as Child-Pugh class A (mild), B (moderate), or C (severe) criteria at screening for Groups 1, 2, or 3, respectively, and documented evidence of hepatic cirrhosis*.

   *by biopsy, nuclear scan, CT, MRI, ultrasound, or other clinically acceptable methods
5. If female, not of childbearing potential* or agrees to avoid becoming pregnant by using acceptable contraception** during the duration of the study.

   *Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral oophorectomy or status after hysterectomy.
   * Females of childbearing potential must agree to use two acceptable methods of contraceptives: bilateral tubal ligation; barrier method (condom) by the male partner (even if vasectomized); hormonal contraceptives; intrauterine contraceptive devices; diaphragm in combination with contraceptive jelly, cream, foam, or spermicide; and abstinence from sexual intercourse with men.
6. If subject is male and capable of reproduction, agrees to avoid fathering a child for three months after dosing by using an acceptable method of birth control*.

   *In addition to the use of a barrier method (condom) even if vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #5, and abstinence from sexual intercourse with women.
7. If the subject is female, a negative serum pregnancy test at screening and a negative urine pregnancy test at admission to the confinement/hospital unit.
8. Willingness to comply with all protocol requirements.

Inclusion Criteria for Non-Hepatically Impaired Controls (Group 4):

1. Subject is able to give voluntary written informed consent before any study related procedure is performed.
2. 18-70 years of age, inclusive.
3. Subject is a healthy volunteer as determined by no clinically significant findings from medical history, physical examination, vital signs, and 12-lead ECG as determined by the Site Investigator.
4. Acceptable laboratory values* obtained at screening (within 21 days prior to admission to the confinement/hospital unit) and either at or within 72 hours of admission to the confinement/hospital unit.

   *Chemistry, complete blood count, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), total bilirubin, alkaline phosphatase, albumin, and urinalysis within the reference range for the test laboratory, unless deemed not clinically significant by the investigator.
5. If female, not of childbearing potential* or agrees to avoid becoming pregnant by using acceptable contraception** during the duration of the study.

   *Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral oophorectomy or status after hysterectomy.

   **Females of childbearing potential must agree to use two acceptable methods of contraceptives: bilateral tubal ligation; barrier method (condom) by the male partner (even if vasectomized); hormonal contraceptives; intrauterine contraceptive devices; diaphragm in combination with contraceptive jelly, cream, foam, or spermicide; and abstinence from sexual intercourse with men.
6. If subject is male and capable of reproduction, agrees to avoid fathering a child for three months after dosing by using an acceptable method of birth control*.

   *In addition to the use of a barrier method (condom) even if vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #5, and abstinence from sexual intercourse with women.
7. If the subject is female, a negative serum pregnancy test at screening and a negative urine pregnancy test at admission to the confinement/hospital unit.
8. Willingness to comply with all protocol requirements.

Exclusion Criteria:

Exclusion Criteria for Patients with Hepatic Impairment (Groups 1-3):

1. Hypokalemia (< 3.5mEq/L), severe hypomagnesemia (< 1.1 mg/dL) or severe hypocalcemia (< 7.5 mg/dL).
2. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 10 times the upper limit of normal.
3. Creatinine clearance < 60 ml/min.
4. Inability to swallow tablets.
5. Presence of any condition or finding* which would jeopardize subject safety, impact study result validity, or diminish the subject's ability to undergo all study procedures and assessments**.

   *in the opinion of the site investigator

   **e.g., inability to draw Pharmacokinetics (PK) samples
6. History of fever or documented fever (oral temperature > / = 100.4 degrees F or > / = 38.0 degrees C) in the 48 hours prior to admission to the the confinement/hospital unit.
7. Currently breastfeeding.
8. History of chronic tobacco/nicotine use (> 10 cigarettes per day for 3 months minimum prior to admission).
9. History of clinically significant allergy or severe side effects with nitroimidazoles (e.g., Metronidazole and related substances and azole antifungals or aromatase inhibitors).
10. Receipt of an investigational drug, vaccine or biologic in a clinical trial within 30 days prior to screening.
11. Use of any over the counter (OTC) medication* within 7 days prior to admission to the confinement/hospital unit, unless** the substance would not likely impact the validity of the study results.

    *including vitamins and herbal supplements, cough and cold medications.

    **in the opinion of the site investigator
12. Treatment with CYP450 enzyme altering drugs* within 7 days prior to admission to the confinement/hospital unit, unless** the substance would not likely impact the validity of the study results.

    * except hormonal contraceptives

      * in the opinion of the site investigator NOTE: See list of CYP450 enzyme altering drugs under the concomitant medications section.
13. A positive blood screen for HIV.
14. A positive alcohol breath test (or other suitable test for alcohol) or a urine screen test for drugs of abuse* at screening and at admission to the confinement/hospital unit.

    *Amphetamines, barbiturates, cocaine metabolites, marijuana, opiates, phencyclidine (PCP).

    NOTE: Results of the urine screen test can be ignored if in the opinion of the PI the results can be explained by the concomitant medications history.
15. Unwillingness to abstain from engaging in strenuous physical activity (e.g. running, bicycling, weightlifting, competitive sports) during the course of the study.
16. Consumption of grapefruit juice in the 48 hours before admission to the confinement/hospital unit, or the inability to abstain from these until completion of Day 12.
17. A Heart Rate-Corrected QT Interval (Fridericia's Formula) (QTcF) interval > 450 msec (males) or > 450 msec (females) at screening (Visit 00A) or admission to the confinement/hospital unit (Visit 00B) or a history of prolonged QTc interval.
18. A family history* of Long QT Syndrome, premature cardiac death**, or sudden death without a preceding diagnosis of a condition*** that could be causative of sudden death.

    *parents

    **due to ischemic heart disease or sudden cardiac death before 55 years of age (men) or 65 years of age (women)

    ***such as known coronary artery disease, congestive heart failure, or terminal cancer
19. Any clinically significant ECG abnormality, in the opinion of the site investigator, at screening and at admission to the confinement/hospital unit.
20. Donation of > 500 mL blood within the 30 days prior to admission to the confinement/hospital unit.
21. Plans to donate blood during the study or up to 14 days after dosing.
22. Persons with a transjugular intrahepatic portosystemic shunt.

Exclusion Criteria for Non-Hepatically Impaired Controls (Group 4):

1. Inability to swallow tablets.
2. Presence of any condition or finding* which would jeopardize subject safety, impact study result validity, or diminish the subject's ability to undergo all study procedures and assessments**.

   *in the opinion of the site investigator

   **e.g., inability to collect Pharmacokinetics (PK) samples
3. History of fever or documented fever (oral temperature > / = 100.4 degrees F or > / = 38.0 degrees C) in the 48 hours prior to admission to the confinement/hospital unit.
4. Currently breastfeeding.
5. History of chronic tobacco/nicotine use (> 10 cigarettes per day for 3 months minimum prior to admission to the confinement/hospital unit).
6. History of seizures (other than febrile seizures during childhood) or known or suspected Central Nervous System (CNS) disorders that may predispose to seizures.
7. History of clinically significant allergy or severe side effects with nitroimidazoles (e.g., Metronidazole and related substances and azole antifungals or aromatase inhibitors).
8. Receipt of an investigational drug, vaccine or biologic in a clinical trial within 30 days prior to screening.
9. Use of any over the counter (OTC) medication* within 7 days prior to admission to the confinement/hospital unit, unless** the substance would not likely impact the validity of the study results.

   *including vitamins and herbal supplements, antacids, cough and cold medications.

   **in the opinion of the site investigator
10. Use of prescription medication except hormonal contraceptives within 30 days prior to admission to the confinement/hospital unit, unless* the substance would not likely impact study result validity.

    *in the opinion of the site investigator
11. Treatment with CYP450 enzyme altering drugs* within 7 days prior to admission to the confinement/hospital unit, unless** the substance would not likely impact the validity of the study results.

    *except hormonal contraceptives

    **in the opinion of the site investigator NOTE: See list of CYP450 enzyme altering drugs under the concomitant medications section.
12. A positive blood screen for HIV.
13. A positive blood screen for hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
14. A positive alcohol breath test (or other suitable test for alcohol) or a urine screen test for drugs of abuse* at screening and at admission to the confinement/hospital unit.

    *Amphetamines, barbiturates, benzodiazepines, cocaine metabolites, marijuana, opiates, phencyclidine (PCP).
15. A history of alcohol abuse or dependence within the past 1 month prior to admission to the confinement/hospital unit.
16. Unwillingness to abstain from engaging in strenuous physical activity (e.g. running, bicycling, weightlifting, competitive sports) during the course of the study.
17. Consumption of grapefruit juice in the 48 hours before admission to the confinement/hospital unit, or the inability to abstain from these until completion of Day 12.
18. A Heart Rate-Corrected QT Interval (Fridericia's Formula) (QTcF) interval > 450 msec (males) or > 450 msec (females) at screening (Visit 00A) or admission to the confinement/hospital unit (Visit 00B) or a history of prolonged QTc interval.
19. A family history* of Long QT Syndrome, premature cardiac death**, or sudden death without a preceding diagnosis of a condition*** that could be causative of sudden death.

    *parents

    **due to ischemic heart disease or sudden cardiac death before 55 years of age (men) or 65 years of age (women)

    ***such as known coronary artery disease, congestive heart failure, or terminal cancer
20. Any clinically significant ECG abnormality, in the opinion of the site investigator, at screening and at admission to the confinement/hospital unit.
21. Donation of > 500 mL of blood within the 30 days prior to admission to the confinement/hospital unit.
22. Plans to donate blood during the study or up to 14 days after dosing.
23. Persons with a transjugular intrahepatic portosystemic shunt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were hepatically impaired or non-hepatically impaired males and females, 18 to 70 years of age, inclusive, and met all eligibility criteria. Enrollment occurred between 29MAR2018 and 22AUG2023.
Groups:
- Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
  PA-824: Pretomanid (PA-824) is a nitroimidazooxazine.
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
  PA-824: Pretomanid (PA-824) is a nitroimidazooxazine.
- Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
  PA-824: Pretomanid (PA-824) is a nitroimidazooxazine.
- Non-hepatically Impaired Controls: Participants with no hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
  PA-824: Pretomanid (PA-824) is a nitroimidazooxazine.
Period: Overall Study
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Started | 6 | 2 | 0 | 6
Completed | 6 | 2 | 0 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the severe hepatic impairment group when the study closed.
Groups:
- Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
- Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
- Non-hepatically Impaired Controls: Participants with no hepatic impairment received a single oral dose of 200mg Pretomanid tablets on day 1
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls | Total
Number analyzed (Participants) | 6 | 2 | 0 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (4.1) | 60.5 (3.5) |  | 59 (7.1) | 60.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 4
  Male | 4 | 1 | 0 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 0 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 4 | 7
  White | 3 | 2 | 0 | 2 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 |  | 6 | 14
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (8.0) | 36.5 (5.0) |  | 27.9 (4.4) | 31.4 (6.3)
Height [Mean (Standard Deviation); unit: cm] | 172.6 (8.2) | 166.4 (12.6) |  | 172.5 (8.6) | 171.7 (8.34)
Weight [Mean (Standard Deviation); unit: kg] | 92.9 (21.8) | 102.4 (29.2) |  | 88.9 (19.5) | 92.5 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-infinity): Area Under the Concentration Time-curve Extrapolated to Infinity at Specified Pre-dose and Post-dose Time Points
Description: AUC(0-infinity) was calculated by noncompartmental analysis using the linear up log down method with the area extrapolated to infinity as Clast/Lambda_z where Clast was the last observed concentration and Lambda_z is the elimination rate constant.
Time Frame: Day 1 to Day 5
Population: The Pharmacokinetics Population consisted of participants in the safety population who had evaluable plasma PK samples for the estimation of Cmax or AUC (0-infinity).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
ng*hr/mL | 34800 (10900) | 55900 (34100) |  | 30700 (6410)

2. Primary Outcome: AUC(0-last): Area Under the Concentration Time-curve to the Last Concentration Above the Lower Limit of Quantitation at Specified Pre-dose and Post-dose Time Points
Description: AUC(0-last) Area under the concentration time-curve to the last concentration above the lower limit of quantitation at specified pre-dose and post-dose time points was calculated by noncompartmental analysis using the linear up log down method.
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
ng*hr/mL | 30800 (9860) | 47500 (26700) |  | 28400 (5130)

3. Primary Outcome: CL/F: Apparent Oral Clearance Calculated From Dose/AUC(0-infinifty) at Specified Pre-dose and Post-dose Time Points
Description: Apparent oral clearance was calculated by noncompartmental analysis using the formula Dose/AUC(0-infinity).
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
L/hr | 6.6 (3.3) | 4.4 (2.7) |  | 6.8 (1.6)

4. Primary Outcome: Cmax: Maximum Pretomanid Concentration at Specified Pre-dose and Post-dose Time Points
Description: Maximum Pretomanid concentration is the maximum observed drug concentration in blood plasma at specified pre-dose and post-dose timepoints.
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
ng/mL | 866 (391) | 1070 (475) |  | 786 (151)

5. Primary Outcome: t(1/2): Apparent Terminal Elimination Half-life at Specified Pre-dose and Post-dose Time Points
Description: Apparent terminal half-life at specified pre-dose and post-dose timepoints was estimated by ln(2)/Lambda_z, where Lambda_z is the elimination rate constant.
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
hr | 29.9 (8.1) | 33.6 (8.1) |  | 23.6 (8.2)

6. Primary Outcome: Tmax: Time of Maximum Pretomanid Concentration at Specified Pre-dose and Post-dose Time Points
Description: Time of maximum Pretomanid concentration (Tmax) at specified pre-dose and post-dose timepoints.
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
hr | 3.2 (1.3) | 7.0 (7.1) |  | 5.7 (2.3)

7. Primary Outcome: Vd/F: Apparent Volume of Distribution at Specified Pre-dose and Post-dose Time Points
Description: Apparent Volume of Distribution at specified pre-dose and post-dose timepoints is the volume that the total amount of administered drug would occupy to provide the same concentration as it currently is in blood plasma divided by the bioavailability. It is calculated by Dose/[Lambda_z x AUC(0-infinity)]
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
L | 280.7 (142.8) | 197.3 (78.5) |  | 222.2 (58.6)

8. Secondary Outcome: Incidence and Severity of Related Adverse Events
Description: Events were determined to be related if there was a reasonable possibility that the study product caused the adverse event (AE); that is, there was evidence to suggest a causal relationship between the study product and the AE. Each event was graded as mild, moderate or severe. Participants are counted according to their maximum severity of the event reported.
Time Frame: Day 1 to Day 12
Population: The Safety Population included all participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
Participants
  Mild | 0 | 0 | 0 | 0
  Moderate | 1 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0

9. Secondary Outcome: Incidence and Severity of Serious Adverse Events
Description: A serious adverse event (SAE) is any adverse event occurring at any dose and regardless of causality that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, is a congenital anomaly or birth defect in an offspring of a subject taking study drug, or is an important medical event.
Time Frame: Day 1 to Day 12
Population: The Safety Population included all participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
Participants
  Mild | 0 | 0 |  | 0
  Moderate | 0 | 0 |  | 0
  Severe | 0 | 0 |  | 0

10. Secondary Outcome: Number of Participants With Abnormal ECG Data
Description: ECG data was collected, including PR interval, QRS duration, QT Interval, QTc interval, RR interval, and Ventricular rate. Abnormal ECG data was evaluated for clinical significance.
Time Frame: Day 12
Population: The Safety Population included all participants who received study product.
Measure: Number; unit: participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
participants
  Clinically Significant | 0 | 0 |  | 0
  Not Clinically Significant | 2 | 0 |  | 2
  No Events Reported | 4 | 0 |  | 4

11. Secondary Outcome: Number of Participants With Abnormal Physical Exam Findings
Description: Summary of physical examination findings were obtained from a comprehensive physical examination including the following body system assessments: skin; head, eyes, ears, nose, and throat; thyroid; neurological; chest and lungs; cardiovascular; abdomen (liver and spleen); lymph nodes; musculoskeletal, and extremities.
Time Frame: Day 3, 4, 5 and 12
Population: The Safety Population included all participants who received study product.
Measure: Number; unit: participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
participants
  Extremities | 0 | 1 |  | 0
  Head, Eyes, Ears, Nose, Throat | 0 | 0 |  | 1
  Musculoskeletal | 1 | 0 |  | 0
  Pulmonary | 1 | 0 |  | 0
  Skin | 2 | 0 |  | 0
  Thyroid | 0 | 0 |  | 0
  Neurological | 0 | 0 |  | 0
  Chest and Lungs | 0 | 0 |  | 0
  Cardiovascular | 0 | 0 |  | 0
  Abdomen (liver and spleen) | 0 | 0 |  | 0
  Lymph Nodes | 0 | 0 |  | 0

12. Secondary Outcome: Number of Participants With Abnormal Safety Laboratory Parameters
Description: Summary of abnormal laboratory parameters were collected following dose of study product through day 12. Abnormal findings were evaluated based on relationship to study product and clinical significance.
Time Frame: Day 2, 5, and 12
Population: The Safety Population included all participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
Participants
  Albumin: Related, Not Clinically Significant | 0 | 0 | 0 | 0
  Albumin: Not Related, Clinically Significant | 0 | 1 | 0 | 0
  Albumin: No Events | 6 | 1 | 0 | 6
  Aspartate Aminotransferase: Related, Not Clinically Significant | 0 | 0 | 0 | 1
  Aspartate Aminotransferase: Not Related, Clinically Significant | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: No Events | 6 | 2 | 0 | 5
  Blood Urea Nitrogen: Related, Not Clinically Significant | 1 | 0 | 0 | 0
  Blood Urea Nitrogen: Not Related, Clinically Significant | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: No Events | 5 | 2 | 0 | 6
  Calcium: Related, Not Clinically Significant | 0 | 0 | 0 | 1
  Calcium: Not Related, Clinically Significant | 0 | 0 | 0 | 0
  Calcium: No Events | 6 | 2 | 0 | 5
  Creatinine: Related, Not Clinically Significant | 0 | 0 | 0 | 1
  Creatinine: Not Related, Clinically Significant | 0 | 1 | 0 | 0
  Creatinine: No Events | 6 | 1 | 0 | 5

13. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs were collected at each study visit following study product administration. Abnormal vital signs were graded as mild, moderate or severe.
Time Frame: Days 1, 2, 3, 4, 5, and 12
Population: The Safety Population included all participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
Number analyzed (Participants) | 6 | 2 | 0 | 6
Participants
  Pulse Rate: Mild | 1 | 0 | 0 | 2
  Pulse Rate: Moderate | 0 | 0 | 0 | 0
  Pulse Rate: Severe | 0 | 0 | 0 | 0
  Pulse Rate: None | 5 | 2 | 0 | 4
  Systolic Blood Pressure: Mild | 1 | 0 | 0 | 1
  Systolic Blood Pressure: Moderate | 0 | 0 | 0 | 0
  Systolic Blood Pressure: Severe | 1 | 0 | 0 | 1
  Systolic Blood Pressure: None | 4 | 2 | 0 | 4
  Diastolic Blood Pressure: Mild | 0 | 0 | 0 | 1
  Diastolic Blood Pressure: Moderate | 1 | 0 | 0 | 1
  Diastolic Blood Pressure: Severe | 1 | 0 | 0 | 0
  Diastolic Blood Pressure: None | 4 | 2 | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first dose of study drug until the final study visit on Day 12.
Description: Within the severe hepatic impairment group, no participants were enrolled prior to study completion.
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Non-hepatically Impaired Controls
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/0 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/0 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 1/2 | 0/0 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=2) | Severe Hepatic Impairment (N=0) | Non-hepatically Impaired Controls (N=6)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02422524/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT02422524/SAP_001.pdf